CLINICAL TRIAL: NCT04357405
Title: Study of the Interest of ECG Teletransmission in Retirement Home (EHPAD) In the Ile-de-France Region.
Acronym: TEECAD
Status: Terminated | Type: Observational
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02647-46
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Pathology; Residents of Retirement Home (EHPAD)
Keywords: ECG; Elderly EHPAD's resident; Cardiac desease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental arm: This group consists of 100 EHPAD which will benefit from ECG teletransmission. all data will be collected
- Control arm: This arm consists of 50 EHPAD that have not benefited from ECG teletransmission. Only the global death occurrence data will be analyzed, no individual data will be collected.

SUMMARY:
The aim of the study is to evaluate the interest and the workability of ECG teletranmission in EHPAD in Île-de-France. ECG for the elderly is beneficial to detect or monitor cardiovascular disease.

DETAILED DESCRIPTION:
Main objectives :

* Evaluate the workability of ECG uploaded by a caregiver who was trained before
* Evaluate the prevalence of ECG anomalies highlighted thanks to the realisation of an uploaded ECG (supraventricular and ventricular rhythm disorder and coronary pathology)

Secondaries objectives :

* Evaluate the prevalence of unknown ECG anomalies and thus determine the number of new diagnostics highlighted thanks to uploaded ECG
* Evaluate the prevalence of ECG iatrogenic anomalies

The study is observational, multicentre and prospective. It is going to include 3211 elderly living in EHPAD in Île-de-France. 150 EHPAD or involved in the study, they are split in two groups : 100 EHPAD will receive ECG and 50 EHPAD will not. This last group will enable to lead a comparative analysis, only global data about death will be collected.

The study will last 36 months with 12 months of participation for each resident.

ELIGIBILITY:
Inclusion Criteria:

Elderly living in nursing homes (EHPAD) who requires electrocadiogram (ECG) due to :

* Cardiac pathology : coronary artery disease, heart failure, high blood pressure, diabetes, valvular disease, atrial fibrillation
* A medication which could causes electrocadiogram (ECG) anomalies Patients living in nursing homes (EHPAD) who give their agreement.

Exclusion criteria :

Protected adult under a protection of the court

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in nursing homes (EHPAD) requiring an electrocadiogram (ECG) except emergency situation, due to a cardiac pathology with / or without treatment which can lead to ECG abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Assessment of teletransmetted electrocardiogram (ECG) feasability (number of ECGs interpretable) | 12 months
  An interpretable ECG is defined by an absence of parasite, a stable baseline, an absence of argument of a malposition of electrodes, an unwinding paper speed: 25 mm / sec, a calibration of the amplitude
Assessment of prevalence of anomalies highlighted by performing an electrocardiogram. | 12 months
  The prevalence of anomalies highlighted by performing an electrocardiogram: supra-ventricular rhythm disorders, ventricular rhythm disorder and coronary pathologies.

SECONDARY OUTCOMES:
Assessment of commorbidity risk and life expectancy according Charlson score. | 12 months
Assessment of prevalence of unknown and iatrogenic anomalies according to the electrocardiogram | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Psychiatric Geriatric Department, Broca hospital
Locations (1):
- Psychiatric Geriatric Department, Broca hospital, Paris, Île-de-France Region, France